CLINICAL TRIAL: NCT02911597
Title: Double-Blind, Cross-Over Trial of Ketamine Therapy Plus or Minus Naltrexone in Treatment Resistant Depression (TRD)
Brief Title: Double-Blind Trial of Ketamine Therapy Plus or Minus Naltrexone in Treatment Resistant Depression (TRD)
Acronym: Ket_Nal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Schatzberg, Alan, M.D. (Individual)
Responsible Party: Principal Investigator, Nolan Williams, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 32105
Record Dates: First submitted 2016-04-23; First posted 2016-09-22 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Depression
Keywords: Ketamine; Naltrexone; Treatment-Resistant; TRD
MeSH Terms: conditions — Depression | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Ketamine + Naltrexone or placebo (Experimental): Patients will receive two infusions of Ketamine 0.5mg/kg divided into two phases Phase A and Phase B, which are separated by 30 days.
  Patients will be randomly assigned to receive either Naltrexone 50 mg or a matched placebo in both Phase A and B. The Naltrexone or placebo will be given 45 min prior to the administration of ketamine 0.5 mg/kg (e.g. patient X assigned to arm X. Arm X is assigned to Ketamine 0.5mg/kg plus Naltrexone 50 mg during Phase A then when transitioning to Phase B they would receive Ketamine 0.5mg/kg plus a matched placebo). In Phase A will then be followed for 30 days with study assessments to examine the durability of Ketamine effects then once at day 30 for transition.
  Interventions: Drug: Naltrexone
- B: Ketamine + Naltrexone or placebo (Experimental): Patients will receive two infusions of Ketamine 0.5mg/kg divided into two phases Phase A and Phase B, which are separated by 30 days.
  Patients will be randomly assigned to receive either Naltrexone 50 mg or a matched placebo in both Phase B and A. The Naltrexone or placebo will be given 45 min prior to the administration of ketamine 0.5 mg/kg (e.g. patient X assigned to arm X. Arm X is assigned to Ketamine 0.5mg/kg plus Naltrexone 50 mg during Phase A then when transitioning to Phase B they would receive Ketamine 0.5mg/kg plus a matched placebo). In Phase B will then be followed for 30 days with study assessments to examine the durability of Ketamine effects then once at day 30 for transition.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — adding naltrexone (or placebo) to a ketamine infusion to potentially block the effects of ketamine as an anti depressant.
  Other Names: Revia

SUMMARY:
The primary objective is to determine if the opioid properties of ketamine are responsible for its antidepressant effects. Since naltrexone can block opiate actions, the investigators will determine if naltrexone can effectively block ketamine's effects.

DETAILED DESCRIPTION:
The primary goal is to determine if the antidepressant effects of Ketamine are mediated by an opiate mechanism.

Primary Objective:

To determine if the opioid properties of Ketamine are responsible for it's antidepressant effects by potentially blocking the antidepressant effects with a opioid antagonist naltrexone.

We will measure this objective by looking at the response on a scale called the 6- item Hamilton Rating Scale for Depression (HAM-D-6). Response is defined as a statistically significant greater decrease on the overall score on this scale, post infusion.

Secondary Objective:

This includes comparing a scale called Clinician Administered Dissociative States Scale (CADSS) on both of our patient groups, one group receiving Ketamine plus Naltrexone compared to the other group receiving Ketamine plus placebeo, to determine if naltrexone has any effect on CADSS as well as to determine if CADSS is associated with antidepressant response

Another secondary objective is to assess ketamine craving using the Visual Analog Craving Scale for Ketamine (VASK), after infusion and determine if there is a change in level of craving for the group that receives naltrexone.

Number of Subjects:

i) 30

ii) The subjects will be drawn from an outpatient sample of patients with MDD, diagnosed with the use of the Structured Clinical Interview for DSM-IV Axis I Disorders(SCID-I/P), currently on a stable, adequate dose of antidepressant therapy, as defined by the MGH ATRQ, for at least 4 weeks or a history of intolerance to at least 2 antidepressant treatments.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion only if all of the following criteria are met:

1. Male or female, 18 to 70 years of age, inclusive, at screening.
2. Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
3. Diagnosed with Major Depressive Disorder (MDD), single or recurrent, and currently experiencing a Major Depressive Episode (MDE) of at least eight weeks in duration, prior to screening, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR™). The diagnosis of MDD will be made by a site psychiatrist and supported by the Structured Clinical Interview for DSM-IV-TR™ (SCID-I/P) or the M.I.N.I International Neuropsychiatric Interview a short, structured psychiatric interview.
4. Has a history of TRD during the current MDE, as assessed by the investigator. TRD is defined as failure to achieve a satisfactory response (e.g., less than 50% improvement of depression symptoms), as perceived by the participant, to at least two "treatment courses" of a therapeutic dose of an antidepressant therapy of at least 8 weeks duration. The adequacy of dose and duration of the antidepressant therapy will be determined as per the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH ATRQ) criteria. Participants must currently be on a stable (for at least 4 weeks) and adequate (according to the MGH ATRQ) dose of ongoing Selective serotonin reuptake inhibitor (SSRI) or Serotonin-norepinephrine reuptake inhibitor (SNRI) antidepressant therapy, of which total duration must be at least 8 weeks. Participants may also have a history of intolerance to at least 2 antidepressant medications. These patients with the intolerance history will not be required to be currently taking an antidepressant medication.
5. Meet the threshold on the total Hamilton Depression 17-item Scale (HAMD17) score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
6. In good general health, as ascertained by medical history, physical examination (PE) (including measurement of supine and standing vital signs), clinical laboratory evaluations, and 12-lead electrocardiogram (ECG).
7. If female, a status of non-childbearing potential or use of an acceptable form of birth control per the following specific criteria:

   1. Non-childbearing potential (e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening); or
   2. Childbearing potential, and meets the following criteria:

   i. Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent.

   ii.Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at randomization prior to receiving study treatment.

   iii.Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.
8. Body mass index between 18-35kg/m2.
9. Concurrent psychotherapy will be allowed if the type (e.g., supportive, cognitive behavioral, insight-oriented, et al) and frequency (e.g., weekly or monthly) of the therapy has been stable for at least three months prior to screening and if the type and frequency of the therapy is expected to remain stable during the course of the subject's participation in the study.
10. Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, or trazodone) will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable during the course of the subject's participation in the study.

Exclusion Criteria:

A potential participant will NOT be eligible for participation in this study if any of the following criteria are met:

1. Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
2. Female that is pregnant or breastfeeding.
3. Female with a positive pregnancy test at screening or baseline.
4. Total HAMD score of <20 at the screen or baseline visits.

6. Current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-IV-TR™), with the exception of nicotine dependence, at screening or within six months prior to screening.

7. Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, or Specific Phobia (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more).

8. History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.

9. History of anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified, within five years of screening.

10. Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within six months prior to screening.

11. Considered at significant risk for suicide during the course of the study according to any of the following criteria:

12. In the judgment of the investigator, the subject is at significant risk for suicidal behavior during the course of his/her participation in the study.

13. Has dementia, delirium, amnestic, or any other cognitive disorder.

14. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results.

15. Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.

16. Known history or current episode of:

a. QTcF (a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle-Fridericia-corrected) ≥450 msec at screening (Visit 1) or randomization b. Syncopal event within the past year. c. Congestive heart failure (CHF) New York Heart Association Criteria >Stage 2 d. Angina pectoris e. Heart rate <50 or >105 beats per minute at screening or randomization

17. Chronic lung disease.

18. Lifetime history of surgical procedures involving the brain or meninges, encephalitis, meningitis, degenerative central nervous system disorder (e.g., Alzheimer's or Parkinson's Disease), epilepsy, mental retardation, or any other disease/procedure/accident/intervention associated with significant injury to or malfunction of the central nervous system (CNS), or a history of significant head trauma within the past two years.

19. Presents with any of the following lab abnormalities w/in the past 6 months:

1. Thyroid stimulating hormone (TSH) outside of the normal limits and clinically significant as determined by the investigator. Free thyroxine (T4) levels may be measured if TSH level is high. Subject will be excluded if T4 level is clinically significant.
2. Any other clinically significant abnormal laboratory result at the time of the screening exam.

   20. History of hypothyroidism and has been on a stable dosage of thyroid replacement medication for less than six months prior to screening.(Subjects on a stable dosage of thyroid replacement medication for at least six months or more prior to screening are eligible for enrollment.)

   21. History of hyperthyroidism which was treated (medically or surgically) less than six months prior to screening.

   22. Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.

   23. History of positive screening urine test for drugs of abuse at screening: cocaine, amphetamines, barbiturates, opiates.

   24. Chronic use of opiates.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Level of Depression as assessed by the HAM-D | Day 1-7
  Compare Hamilton of Naltrexone versus Placebo administered during ketamine infusion for depression.

SECONDARY OUTCOMES:
Level of Depression as assessed by the Beck Depression Inventory (BDI) | Day 1-7
  Compare Beck of Naltrexone versus Placebo administered during ketamine infusion for depression.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schatzberg, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Williams NR, Heifets BD, Blasey C, Sudheimer K, Pannu J, Pankow H, Hawkins J, Birnbaum J, Lyons DM, Rodriguez CI, Schatzberg AF. Attenuation of Antidepressant Effects of Ketamine by Opioid Receptor Antagonism. Am J Psychiatry. 2018 Dec 1;175(12):1205-1215. doi: 10.1176/appi.ajp.2018.18020138. Epub 2018 Aug 29. PMID 30153752